CLINICAL TRIAL: NCT00209820
Title: Nordic Walking and Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Human Locomotion Science (Other)
Collaborators: Nordic Institute of Chiropractic and Clinical Biomechanics (Other); University of Southern Denmark (Other); Hospitals of Funen (Unknown); National Board of Health, Denmark (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: VF 20050055
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2005-09

CONDITIONS: Low Back Pain
Keywords: low back pain; randomized clinical trial; Nordic walking; supervision; Advice to stay active
MeSH Terms: conditions — Low Back Pain

INTERVENTIONS:
Behavioral: Supervised Nordic Walking
Behavioral: Unsupervised Nordic Walking
Behavioral: Advice to stay active

SUMMARY:
This is a randimized clinical trial comparing the effect of supervised Nordic walking versus unsupervised Nordic walking versus advice to stay active

ELIGIBILITY:
Inclusion Criteria:

* Finished treatment at secondary sector specialist spinal unit
* Able to understand and read Danish

Exclusion Criteria:

* Co-morbidity preventing patient from completing Nordic walking program
* Pain <3 on 11 point box scale
* Unable to perform Watt Max Cykel Test

Ages: 8 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150
Dates: Start 2005-09; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Morsø, PT, Study Director — Back Center Funen, Ringe Denmark; Jan Hartvigsen, DC, PhD, Principal Investigator — Nordic Institute of Chiropractic and Clinical Biomechanics; Claus Manniche, MD, PhD, Study Chair — Back Center Funen, Ringe, Denmark
Locations (1):
- Back Center Funen, Ringe, Funen, Denmark

REFERENCES:
- [Background] Morso L, Hartvigsen J, Puggaard L, Manniche C. Nordic walking and chronic low back pain: design of a randomized clinical trial. BMC Musculoskelet Disord. 2006 Oct 2;7:77. doi: 10.1186/1471-2474-7-77. PMID 17014731
- [Derived] Hartvigsen J, Morso L, Bendix T, Manniche C. Supervised and non-supervised Nordic walking in the treatment of chronic low back pain: a single blind randomized clinical trial. BMC Musculoskelet Disord. 2010 Feb 10;11:30. doi: 10.1186/1471-2474-11-30. PMID 20146793